CLINICAL TRIAL: NCT03511339
Title: Pro-2-Cool Device Clinical Study: an Assessment of Clinical Efficacy of Hypothermic Therapy Following Mild Traumatic Brain Injury (mTBI) in the Adolescent Athlete as Compared to an Untreated Active Control Population
Brief Title: Pro-2-Cool Device Clinical Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TecTraum Inc. (Industry)
Collaborators: Bright Research Partners (Industry); Akron Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1289670
Record Dates: First submitted 2018-03-30; First posted 2018-04-27 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-05

CONDITIONS: Mild Traumatic Brain Injury
Keywords: Concussion; TBI; mTBI
MeSH Terms: conditions — Brain Concussion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Control (No Intervention): Brain rest
- TecTraum Device (Experimental): Treatment with study device
  Interventions: Device: TecTraum device

INTERVENTIONS:
Device: TecTraum device — A non-invasive hypothermic therapy ("cold therapy") TecTraum device that provides localized cooling of the head and neck.
  Other Names: Pro-2-Cool
  Arms: TecTraum Device

SUMMARY:
This study is being conducted to quantify the clinical safety and efficacy of head and neck cooling when applied up to 8 days after mild traumatic brain injury (mTBI) among adolescents participating in sporting activities.

DETAILED DESCRIPTION:
This is a single-center, prospective, randomized, non-blinded, dual-arm comparator study that will include two-phases, the 60-patient pilot study (30 patients in the treatment arm and 30 patients in the control arm) followed by a pivotal study (up to 200 patients in the treatment and control arm combined) for a total of up to 260 patients overall in both phases. The pilot study will serve as an opportunity to assess the protocol and make adjustments, if necessary. In addition, descriptive statistics including effect size will be calculated and the safety of the device will be assessed at the conclusion of the pilot study.

Subjects will be assigned to study arm based on a block randomization schedule generated a priori.

The study sponsor believes that the device and therapeutic treatment that will be evaluated in this study is a non-significant risk (NSR) to the subjects.

ELIGIBILITY:
Inclusion Criteria:

* Males and females ages 12 - 21 years
* Initial provider visit is within 8 days of mTBI injury
* Confirmed mTBI diagnosis from sporting activities
* In generally good health as confirmed by medical history and as determined by site investigator
* Has a symptom score of at least 7 (analogous of the SCAT5 symptoms score)
* Has informed consent obtained per protocol and as required per Institutional Review Board (IRB)

Exclusion Criteria:

* Cleared to return to play during initial visit
* Suffers a serious TBI as evidenced by worsening symptoms, specifically:
* Seizure
* Hospitalization
* Existing positive diagnostic testing, which include radiology scans that indicate brain bleed
* Slurred speech, which has not resolved within 72 hours of mTBI injury
* Sustains another head or neck injury at the time of mTBI injury which requires medical treatment
* Known or disclosed pregnancy or breast-feeding
* History of a serious medical or psychiatric disorder that include:

  * Suicide attempt in the last 6 months
  * Unmanaged depression or anxiety
  * Hospitalization in the last 6 months for psychiatric treatment
* History of Reynaud's disease or phenomenon, cold agglutinin disease, cryoglobulinemia, or cryofibrinogenemia
* Previously diagnosed with a cerebrovascular disorder
* Is unable to understand the study requirements or the informed consent
* Currently enrolled in another investigational research study that may confound the results of this study
* Non-English speaking subjects and parents/legal guardians

Ages: 12 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 174 (Actual)
Dates: Start 2017-11-04 (Actual); Primary Completion 2022-04-27 (Actual); Study Completion 2022-05-29 (Actual)

PRIMARY OUTCOMES:
The SCAT5 overall score will be collected at the initial visit in the Sports Medicine Clinic, and compared to follow-up visits throughout the study, with the objective of demonstrating better outcomes in the treatment group compared to the control group. | Change from initial visit to 4 weeks
  Formal statistical hypothesis testing will be employed in the evaluation of this endpoint.
  Additionally, comparisons between treatment groups on the baseline SCAT5 (SCAT5-PRE) will be performed at initial visit (as reported by subject) and at each follow-up (72 hours, 10 days, and 4 weeks) separately to evaluate the time trend in recovery. Individual SCAT5 symptoms, each scored on a scale of 0-6, will also be summarized and compared by treatment group to investigate the effect of treatment on specific symptoms. These comparisons are intended to provide additional information on the pattern of recovery and are not attached to intended labeling claims; however, statistical testing of these endpoints will be accompanied by adjustment for multiplicity using the Hochberg-Holm method.

SECONDARY OUTCOMES:
Recovery time from initial visit, summarized by group and compared in the treatment group to control. | Initial visit through earliest follow up where complete recovery is observed, maximum of 4 weeks after initial visit.
  Recovery time from initial visit will be formally evaluated for differences between treatment and control.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Congeni, MD, Principal Investigator — Akron Children's Hospital
Locations (5):
- United States (5):
  - University of Michigan - Michigan Medicine, Ann Arbor, Michigan
  - Akron Children's Hospital, Akron, Ohio
  - Akron Children's Hospital, Mahoning Valley Campus, Boardman, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Dayton Children's Hospital, Dayton, Ohio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Congeni J, Murray T, Kline P, Bouhenni R, Morgan D, Liebig C, Lesak A, McNinch NL. Preliminary Safety and Efficacy of Head and Neck Cooling Therapy After Concussion in Adolescent Athletes: A Randomized Pilot Trial. Clin J Sport Med. 2022 Jul 1;32(4):341-347. doi: 10.1097/JSM.0000000000000916. Epub 2021 Mar 10. PMID 34009790
- See also: TecTraum website with video describing trial. — https://www.pro-2-cool.com/